CLINICAL TRIAL: NCT05222464
Title: Utilizing MyChart to Assess the Effectiveness of Interventions for Vasomotor Symptoms: A Feasibility Study (REaCT-Hot Flashes Pilot)
Brief Title: Utilizing MyChart to Assess the Effectiveness of Interventions for Vasomotor Symptoms: A Feasibility Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REaCT-Hot Flashes Pilot
Record Dates: First submitted 2021-12-15; First posted 2022-02-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Vasomotor Symptoms; Machine Learning
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of Care Intervention (Other): Standard of care intervention - The intervention will consist of 4 classes of standard of care treatments, namely, lifestyle modifications, complementary and alternative medicine (CAM) therapies, prescription medications, or adjustment of anti-cancer therapy.
  Interventions: Other: Standard of care treatments

INTERVENTIONS:
Other: Standard of care treatments — Interventions will consist of 4 classes of standard of care treatments, namely, lifestyle modifications, complementary and alternative medicine (CAM) therapies, prescription medications, or adjustment of anti-cancer therapy.

SUMMARY:
Vasomotor symptoms (VMS) are a common consequence of systemic therapies for breast cancer. Breast cancer treatments can cause VMS in approximately 30% of postmenopausal women and 95% of premenopausal women with early stage breast cancer (EBC). There are many non-estrogen-based interventions available to manage VMS, including; lifestyle modifications, complementary and alternative medicine (CAM) therapies. However, a recent systematic review and meta-analysis of pharmacological and CAM interventions conducted by our team, found no single optimal treatment for VMS management in breast cancer patients. Given the complex patient, cancer and treatment variables influencing the experience of VMS, the numerous potentially effective VMS interventions available and the varying expectations for an effective intervention, the investigators believe Machine Learning (ML) is ideally suited to the analysis of this common and bothersome treatment related toxicity. The EPIC electronic medical record, and MyChart application has provided both clinicians and patients with increased tools for the documentation of health related outcomes. The investigators believe that the MyChart platform, and ML techniques can be utilized to collect, and analyze outcome data for breast cancer patients experiencing VMS.

DETAILED DESCRIPTION:
Vasomotor symptoms (VMS) are a common consequence of systemic therapies for breast cancer. Breast cancer treatments can cause VMS in approximately 30% of postmenopausal women and 95% of premenopausal women with early stage breast cancer (EBC). In addition to their negative impact on quality of life, unmanaged VMS are the most common reason for discontinuation of potentially curative treatment in 25-60% of EBC patients. Estrogen replacement is a common treatment for VMS in the general population, however, it is contraindicated in breast cancer patients. There are many non-estrogen-based interventions available to manage VMS, including; lifestyle modifications, complementary and alternative medicine (CAM) therapies. However, a recent systematic review and meta-analysis of pharmacological and CAM interventions conducted by our team, found no single optimal treatment for VMS management in breast cancer patients. The investigators recently conducted a survey in 373 patients with EBC which found that while the majority of patients were interested in receiving an intervention to mitigate their symptoms, only 18% received a treatment for this problem. In addition, more than one third of patients experiencing VMS report that they are not routinely asked about their symptoms in routine follow up. Given the complex patient, cancer and treatment variables influencing the experience of VMS, the numerous potentially effective VMS interventions available and the varying expectations for an effective intervention, the investigators believe Machine Learning (ML) is ideally suited to the analysis of this common and bothersome treatment related toxicity. Prior breast cancer studies have successfully applied to ML models to examine risk of developing breast cancer, as well as breast cancer prognosis. The EPIC electronic medical record, and MyChart application has provided both clinicians and patients with increased tools for the documentation of health related outcomes. The investigators believe that the MyChart platform, and ML techniques can be utilized to collect, and analyze outcome data for breast cancer patients experiencing VMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who have histologically confirmed breast cancer, of any stage
* Patients experiencing vasomotor symptoms
* While the study is intended to evaluate the feasibility of the MyChart platform, patients without a MyChart account, who are interested in participating in the study, will have access to a paper or electronic email version. As participation in the MyChart program has benefits outside of this intended study, all patients without a MyChart account will be encouraged to sign up for the service

Exclusion Criteria:

* Those who are unable to complete questionnaires in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Patient Engagement (MyChart Accessibility and User Experience) | 3 Months
  Patient engagement will be defined by 60% of patients approached agreeing to participate in the study.
Physician Engagement (MyChart Accessibility and User Experience) | 3 Months
  Physician engagement will be defined by 60% of those completing the study log to approach patients for participation in study.
Patient Accrual (MyChart Accessibility and User Experience) | 3 Months
  Patient accrual will be defined by accruing 50 participants within 3 months.
MyChart Utilization | Baseline and 6 weeks
  MyChart utilization will be defined as 85% of participants completing both questionnaires (the Hot Flash Problem Score and the Composite Hot Flash Score) on the MyChart interface, and 50% of enrolled participants completing both questionnaires as per study protocol.

SECONDARY OUTCOMES:
Hot Flash Severity (MyChart Feasibility) | 3 Months
  Hot flash severity (MyChart feasibility) will be assessed by the Hot Flash Problem Score, a composite score of the perceived distress, interference, and problematic nature of vasomotor symptoms (VMS) in daily life and by the composite hot flash score (assess hot flashes on a daily basis for 7 days). The researchers will assess the feasibility of using MyChart to complete hot flash severity assessments by determining the percentage of participants who complete the tools as per protocol, including the percentage of patients who complete daily assessments over the 7 day period.
MyChart Feasibility in assessing effectiveness of interventions for VMS | 3 months
  The investigators will assess the effectiveness of an intervention by assessing change in hot flash severity scores using the Hot Flash Problem Score, and composite hot flash score from baseline to 6 weeks post intervention.
Effectiveness of Interventions for VMS - Traditional Statistical Modeling | 3 Months
  Analyze MyChart questionnaire response data, using traditional statistical modelling (including linear and logistic regression models) to predict change in hot flash severity outcomes in response to interventions for VMS. The severity outcomes will be based on two validated clinical tools. These tools consist of the Hot Flash Problem Score (a composite score of the perceived distress, interference, and problematic nature of VMS in daily life), and Composite Hot Flash Score (this assess hot flashes on a daily basis for 7 days).
Effectiveness of interventions for VMS (MyChart feasibility) | 3 Months
  Effectiveness of interventions for VMS (MyChart feasibility) will be assessed by frequency of nocturnal awakenings, and toxicity data. Data will be analyzed using traditional statistics and machine learning techniques to create a preliminary model predicting VMS treatment response in individuals.
Predicting effectiveness of interventions for VMS - machine learning | 3 Months
  Utilize machine learning models, including classification and regression trees, with comparison against standard regression models, to assess for improvements in predictive power for hot flash severity. The researchers will use model explainability techniques, such as conditional dependence plots, to study the impact of specific features on the hot flash severity outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McGee, MD, Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Cole KM, Clemons M, McGee S, Alzahrani M, Larocque G, MacDonald F, Liu M, Pond GR, Mosquera L, Vandermeer L, Hutton B, Piper A, Fernandes R, Emam KE. Using machine learning to predict individual patient toxicities from cancer treatments. Support Care Cancer. 2022 Sep;30(9):7397-7406. doi: 10.1007/s00520-022-07156-6. Epub 2022 May 25. PMID 35614153
- [Background] Hutton B, Hersi M, Cheng W, Pratt M, Barbeau P, Mazzarello S, Ahmadzai N, Skidmore B, Morgan SC, Bordeleau L, Ginex PK, Sadeghirad B, Morgan RL, Cole KM, Clemons M. Comparing Interventions for Management of Hot Flashes in Patients With Breast and Prostate Cancer: A Systematic Review With Meta-Analyses. Oncol Nurs Forum. 2020 Jul 1;47(4):E86-E106. doi: 10.1188/20.ONF.E86-E106. PMID 32555553
- [Background] Cole KM, Clemons M, Alzahrani M, Larocque G, MacDonald F, Vandermeer L, Hutton B, Piper A, Pond G, McGee S. Developing patient-centred strategies to optimize the management of vasomotor symptoms in breast cancer patients: a survey of health care providers. Breast Cancer Res Treat. 2021 Jul;188(2):343-350. doi: 10.1007/s10549-021-06186-8. Epub 2021 Jun 22. PMID 34159473
- [Result] Cole KM, McGee S, Clemons M, Liu M, MacDonald F, Vandermeer L, Ng TL, Pond G, Emam KE. Development and application of a weighted change score to evaluate interventions for vasomotor symptoms in patients with breast cancer using regression trees: a cohort study. Breast Cancer Res Treat. 2024 Sep;207(2):313-321. doi: 10.1007/s10549-024-07360-4. Epub 2024 May 19. PMID 38763972
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/